CLINICAL TRIAL: NCT02034474
Title: Tocilizumab, An IL-6 Receptor Antibody, As Add-On Treatment For Residual Positive, Negative, and Cognitive Symptoms of Schizophrenia: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Tocilizumab as Add-On Treatment For Residual Positive, Negative, and Cognitive Symptoms of Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Marlene Carlson, Assistant Professor of Psychiatry at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6729
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tocilizumab (Experimental): Tocilizumab will be administered at day 0, week 4 and week 8 via an iv drip over 60 min. Dose is 8mg/kg but may be reduced to 4mg/kg if intolerable. Maximum dose will be 800mg.
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): Placebo will be administered intravenously via an iv drip over 60 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — 8mg/kg intravenously via iv drip over 60 min
  Other Names: Actemra
  Arms: tocilizumab
Drug: Placebo — intravenously via iv drip over 60 min
  Other Names: Saline Drip
  Arms: Placebo

SUMMARY:
Randomized, double-blind clinical trial of tocilizumab vs. placebo as add-on treatment for residual positive, negative, and cognitive symptoms in schizophrenia. The primary study hypothesis is that individuals receiving tocilizumab will show greater improvements in their PANSS total scores than those taking placebo.

DETAILED DESCRIPTION:
One of the main mediators of the effects of infection/inflammation in the human body is cytokines. Recent data suggest that cytokines, and in particular IL-6, may mediate the effects of lifetime or prenatal infection on schizophrenia risk. Preclinical models of schizophrenia support a convergence between a role for IL-6 in the pathophysiology of schizophrenia and the major neurochemical hypotheses of schizophrenia-the dopamine and glutamate hypotheses. Namely, IL-6 dysfunction or excess promotes schizophrenia-like behaviors and schizophrenia-like biochemical and electrophysiological profiles, while IL-6 knockout or neutralization mitigates these abnormalities. Furthermore, plasma IL-6 levels are elevated in acutely psychotic but not treated patients, and Positron Emission Tomography (PET) studies have shown active inflammation in the brains of individuals with psychosis. Finally, treatment of individuals with schizophrenia with non-specific anti-inflammatory agents, such as celecoxib and aspirin, has suggested a role for anti-inflammatory agents in schizophrenia. These data also suggest that studies of immunologic agents that more specifically target the underlying pathophysiology of schizophrenia may be more efficacious. Tocilizumab (Actemra®) is an FDA-approved humanized monoclonal antibody against the IL-6 receptor used for treatment of rheumatoid arthritis in individuals who have not responded to at least one TNF-alpha therapy and for juvenile idiopathic arthritis

ELIGIBILITY:
Inclusion Criteria:

* Fulfill DSM-IV criteria for schizophrenic illness, schizoaffective disorder
* Negative urine toxicology
* Capacity to understand the study and give written informed consent
* Must be on a stable dose of antipsychotic medications, up to two medications, except for clozapine, for at least 4 weeks if oral or 2 cycles if depot. Mood stabilizers, benzodiazepines and antidepressants are allowed as long as no change for 4 weeks.
* Moderate level of symptomatology

Exclusion Criteria:

* Pregnancy or lactation, lack of effective birth control during the 15 days before the initial day of the study and for the duration of the drug trial
* Unstable medical or neurological condition (including chronic rashes other than mild eczema, ANC < 2000, platelet count < 120,000, severe liver disease or AST/ALT greater than 1.5 times the ULN at baseline, or any chronic inflammatory or immunologic disorder that impairs the immune system, a current severe infection, intestinal diverticula, or tuberculosis (latent or active-patients with a positive ppd but negative chest x ray may participate) or a live vaccine within one month of receiving study drug
* Any current non medicinal use of amphetamines, opiates, cocaine, sedative-hypnotics, cannabis, or other psychoactive drugs (other than nicotine)
* Currently taking a medication known to cause neutropenia (clozapine, carbamazepine), or another disease modifying anti-rheumatic drugs (DMARD)
* Any history of substance dependence (other than nicotine or cannabis) within the previous 6 months or a history of substance abuse within the previous 1 month (other than nicotine)
* Impaired intellectual functioning
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer)
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples are CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline
* Previous treatment with tocilizumab (an exception to this criterion may be granted for single dose exposure upon application to the sponsor on case-by-case basis
* Any previous treatment with alkylating agents such as chlorambucil, or with a total lymphoid irradiation
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease)
* Current liver disease
* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, Hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks or oral antibiotics within 2 weeks
* Active TB requiring treatment within the previous 3 years.
* Primary or secondary immunodeficiency (history of or currently active)
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured) or breast cancer diagnosed within the previous 20 years
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation
* Lack of peripheral venous access
* Body weight of >150 kg
* Serum creatinine > 1/6mg/dL (141 umol/L) in female patients and > 1.9 mg/dL (168 umol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study if their estimated glomerular filtration rates (GFR) are > 30
* Total Bilirubin >ULN
* Hemoglobin < 85g/L
* White Blood Cells <3.0 x 10^9/L
* Absolute Lymphocyte Count < 0.5 x 10^9/L
* Positive Hepatitis BsAg or Hepatitis C antibody

Additional Exclusion Criteria for MRI portion

* Metal implants or a history of metal working
* Lifetime diagnosis of asthma with asthmatic symptoms within the past 3 years
* Lifetime diagnosis of renal failure or renal disease
* Lifetime diagnosis of hypertension or diabetes
* Renal insufficiency
* More than one previous gadolinium scan

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ragy R Girgis, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 59 subjects who signed consent, 22 did not receive study drug. In addition, one of the 37 subjects who received study drug did not participate in any follow up assessments so was not included in the ITT analysis
Groups:
- Tocilizumab: Tocilizumab (N=19)
- Placebo: Placebo (N=17)
Period: Overall Study
Arm/Group | Tocilizumab | Placebo
Started | 19 | 17
1 Dose | 2 | 4
2 Doses | 2 | 0
3 Doses | 15 | 13
Completed | 15 | 13
Not Completed | 4 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Population: One subject was randomized but received no follow up study assessments so was not included in the ITT analysis
Groups:
- Placebo: Placebo-receiving group
- Tocilizumab: Tocilizumab-receiving group
- Total: Total of all reporting groups
Arm/Group | Placebo | Tocilizumab | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: ITT population
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 19 | 36
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: yrs] — Population: ITT Population
  yrs | 41.67 (10.25) | 43.24 (11.42) | 42.50 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Female | 4 | 7 | 11
    Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Hispanic or Latino | 1 | 5 | 6
    Not Hispanic or Latino | 16 | 14 | 30
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 6 | 12 | 18
    White | 9 | 5 | 14
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    United States | 17 | 19 | 36
PANSS Total [Mean (Standard Deviation); unit: panss score] — Positive and Negative Symptom Scale, Total Score (Sum of all subscales) Minimum = 30, Maximum = 210 Higher score = greater symptomatology
  panss score | 73.94 (15.52) | 70.68 (11.2) | 72.22 (14.24)
Smoker [Count of Participants; unit: Participants] | 7 | 8 | 15
cigs /day [Mean (Standard Deviation); unit: cigarettes per day] | 8 (3) | 10 (5) | 9 (4)
chlorpromazine equivalents [Mean (Standard Deviation); unit: milligrams] — Dosages of antipsychotic medications for each individual were converted to corresponding equivalent dose of chlorpromazine, in milligrams Population: Some participants did not provide antipsychotic dosage information to be converted to chlorpromazine equivalent
  milligrams
    number analyzed (Participants) | 12 | 5 | 17
    (all) | 377 (346) | 257 (192) | 310 (396)
weight [Mean (Standard Deviation); unit: pounds] | 203.24 (51.95) | 218.63 (45.24) | 211.36 (44.01)
Clinical Global Impression - Severity Scale [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated severity of illness
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
  units on a scale | 4 (0.4) | 4 (0.3) | 4 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Tocilizumab
Description: To evaluate an anticipated clinical response to tocilizumab treatment including positive, negative and cognitive symptoms by the change in the Positive and Negative Syndrome Scale (PANSS) total score. Score ranges from 30 to 210 for PANSS total, 16-112 for General, 7-49 for positive and 7-49 for negative symptoms subscales. A lower score means less symptomatic. There is a total score and general psychopathology scores, a positive symptoms score and a negative symptom score. The unit of measure is units on a scale from 1-7, whole numbers only. Summed scores are simply added to each other
Time Frame: Baseline (start of tocilizumab) through 12 weeks. We present the change scores
Population: 17 placebo patients and 19 tocilizumab patients were included in the ITT analysis
Measure: Mean (Standard Deviation); unit: Units on a scale (PANSS)
Groups:
- Placebo: Patients on placebo
- Tocilizumab: Patients on Tocilizumab
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 17 | 19
Units on a scale (PANSS) | -5.33 (17.96) | -0.5 (12.62)

2. Secondary Outcome: Cognitive Symptomatology - Overall MATRICS t Score Change
Description: MATRICS cognitive consensus battery, overall t score change. The composite T-score at each time point (baseline and week 12) is a T-Score (ranging from 0 to 100) reflecting overall neuropsychological function, aggregated from the participant's T-scores on the MATRICS subscales for Speed of Processing, Attention/Vigilance, Working Memory, Verbal Learning, Visual Learning, Reasoning and Problem Solving, and Social Cognition. The outcome is the difference between overall composite T-score at baseline and week 12, with higher difference score reflecting a greater improvement in neuropsychological performance.
Time Frame: Baseline (start of tocilizumab) through 12 weeks
Population: These subjects were included in the ITT analysis and received the MATRICS. We will present total composite change scores from baseline to week 12
Measure: Mean (Standard Deviation); unit: T Score Difference
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 17 | 19
T Score Difference | 2.83 (5.59) | 1.47 (8.53)

3. Secondary Outcome: Cognitive Symptomatology - UPSA-B Score Change
Description: At Baseline and Week 12, participants are UPSA-B given items reflecting ability to complete tasks encountered in daily life, across two domains, Financial Skills and Communication Skills. % correct is calculated for each domain and converted to a standardized score from 0-50. These scores are summed to produce a total summary score ranging from 0-100. The outcome is the difference between this summary score at Baseline and Week 12, with a higher difference score reflecting a greater increase in functional capacity.
Time Frame: Baseline (start of tocilizumab) through 12 weeks
Population: These subjects were included in the ITT analysis and received the UPSA at both baseline and week 12.We will present total composite change scores from baseline to week 12
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 16 | 12
Change in score on a scale | 1.12 (0.23) | 1.12 (0.17)

4. Other Pre Specified Outcome: Relationship Between Baseline IL-6 Levels and Positive, Negative and Cognitive Symptoms and Impairment
Description: Comparison of cytokines, in particular IL-6 levels and the positive, negative and cognitive symptoms and impairments in daily functioning in schizophrenia. These outcomes will be measured by Positive and Negative Syndrome Scale (PANSS), Global Assessment of Functioning (GAF), Clinical Global Impression (CGI), University of California Performance Skills Assessments (UPSA) and MATRICS.
Time Frame: Baseline (start of tocilizumab) through 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Placebo: Subjects who received placebo
- Tocilizumab: Subjects who received tocilizumab
Arm/Group | Placebo | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/19
Other Adverse Events (participants affected / at risk) | 4/17 | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Tocilizumab (N=19)
agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Tocilizumab (N=19)
Inpatient admission (Nervous system disorders) | 1 (1) | 1 (1) — Psychiatric Decompensation
Low ANC (Blood and lymphatic system disorders) | 2 (2) | 2 (2) — ANC between 1000-2000 cells/ul
URI (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — upper respiratory tract infection
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) — tooth infection
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — nausea
fatigue (General disorders) | 0 (0) | 1 (1) — fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT02034474/Prot_000.pdf
  • Informed Consent Form (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02034474/ICF_001.pdf
  • Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02034474/SAP_002.pdf